CLINICAL TRIAL: NCT04543799
Title: SIESTA: A Pilot Observational Study to Investigate and Evaluate Sleep Quality in Cancer Patients Undergoing Hormonal Therapeutic Approaches: 1) Localized, Locally Advanced or Metastatic Prostate Cancer Receiving Treatment Including Androgen Deprivation Therapy 2) Full-resected Early (Stage I-III) Breast Cancer, Ductal Carcinoma in Situ or Lobular Carcinoma in Situ, Without Evidence of Residual Disease; Proven Postmenopausal Status
Brief Title: Evaluation of Sleep Quality in Prostate Cancer Patients Undergoing Treatment With Hormonal Therapeutic Approaches and in Patients With Full-resected Early Breast Cancer
Acronym: SIESTA
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: SIESTA_01
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms | interventions — Polysomnography; Actigraphy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A1: Group A1 consists of patients with prostate cancer receiving ADT as part of their standard care for either locally advanced or metastatic disease.
  Group A1 consists of a combination of two groups; B1, metastatic patients receiving ADT both with and without an oral AR targeted agent, and not receiving radiotherapy and B2, locally advanced patients receiving ADT alongside radiotherapy
  Interventions: Device: polysomnography, actigraphy, questionnaires
- A2: patients with localised prostate cancer receiving radiotherapy only
  Interventions: Device: polysomnography, actigraphy, questionnaires
- YET: Breast cancer survivors receiving endocrine therapy
  Interventions: Device: polysomnography, actigraphy, questionnaires
- NET: Breast cancer survivors not receiving endocrine therapy
  Interventions: Device: polysomnography, actigraphy, questionnaires

INTERVENTIONS:
Device: polysomnography, actigraphy, questionnaires — sleep quality recording

SUMMARY:
This study will use polysomnography, alongside other methodologies such as questionnaires, actigraphic measurements and salivary melatonin samples used in previous studies to investigate sleep quality in patients with i) localized, locally advanced or metastatic hormone sensitive prostate cancer or ii) with full-resected early (stage I-III) epithelial breast cancer. The measurements will be taken before androgen deprivation therapy (ADT - for prostate cancer patients) or endocrine therapy (for breast cancer patients) is initiated, at 6 months and some measures again at 12 months.The groups, defined by cancer type and whether or not treatment includes ADT / endocrine therapy, will be compared to see if there are differences in the prevalence of the lowered sleep quality in the groups.

DETAILED DESCRIPTION:
The main outcomes of this pilot study can be summarised as:

* Using a previously unused methodology to assess whether ADT / endocrine therapy may negatively affect patterns of sleep quality
* Identifying sleep micro/macrostructure changes in prostate cancer patients receiving ADT / endocrine therapy
* Comparing the novel methodology with results obtained previously through standard methods
* Providing statistical underpinnings, such as sample size calculations, for a full interventional trial
* Highlighting the most appropriate non-pharmaceutical interventions to be tested in the full interventional trial

ELIGIBILITY:
Inclusion Criteria for prostate cancer patients:

* Written infor med consent according to International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) regulations before registration and prior to any trial specific procedures
* Histologically proven adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group performance status 0-2
* Adult male patient > 18 years of age, no upper age limit
* Localized prostate cancer, locally advanced hormone-sensitive prostate cancer (HSPC) or metastatic hormone-sensitive prostate cancer (mHSPC)
* ADT recipients are required to be scheduled to start ADT as standard of care (SOC) for metastatic or locally advanced prostate cancer
* Scheduled to receive ADT treatment as SOC for > 6 months in combination with radiotherapy or oral AR-targeted systemic treatment as prescribed by the treating physician or radiotherapy alone

Exclusion Criteria for prostate cancer patients:

* Histology with predominant small cell prostate cancer
* Any previous treatment with ADT or oral AR-targeted agent (exception for short course anti-androgens - disease flare)
* Have not received systemic treatment for any other cancer within the last 12 months
* Active secondary malignancy that requires systemic therapy
* Any clear contraindications present against treatment with ADT
* Presence of sleep apnea syndrome, Apnea Hypopnea Index (AHI) >15 at baseline
* Body mass index (BMI) > 35 at baseline
* Severe respiratory disorders (asthma, Chronic obstructive pulmonary disease) at baseline
* Severe cardiovascular disease or severe cardiovascular event < 6 months
* History of stroke or other neurologic chronic illnesses < 6 months
* Have demonstrated impaired mental status
* History of brain tumours, presence of brain metastases or previous cranial irradiation
* Night shift workers
* Excessive lifestyle: massive coffee intake at night, regular excessive cigarette and alcohol consumption in the evening
* Unhealthy sleep hygiene
* Nocturia (the urgent need to urinate more than 2 times during the main sleep period at night) at baseline
* Present diagnosis of depression or psychiatric illness pharmacologically treated
* Diagnosis of insomnia and chronic intake of hypnotic medication at baseline
* Chronic intake of medications that are known to induce sleep disturbance (antihistamines of first generation, cortisone intake > 25 mg/day)
* Any diagnosed condition that causes known sleep disturbance

Inclusion criteria for breast cancer patients

* Written informed consent according to International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) regulations before registration and prior to any trial specific procedures
* Women with full-resected early (stage I-III) epithelial BC, ductal carcinoma in situ or lobular carcinoma in situ, without evidence of residual disease
* Eastern Cooperative Oncology Group performance status 0-2
* Adult female patient ≥ 18 years of age, no upper age limit
* Proven postmenopausal status (defined by absence of menstruation for at least 6 months and/or level of estradiol <40 pg/ml, or bilateral oophorectomy or ovarian irradiation for suppression of ovarian function)

Exclusion criteria for breast cancer patients

* Non-epithelial BC or BC with mixed epithelial and non-epithelial histology
* Previous chemotherapy at any time, in treatment with ET at not standard dosage
* Have received systemic treatment for any other cancer within the last 12 months
* Active secondary malignancy that requires systemic therapy
* Presence of sleep apnea syndrome, Apnea Hypopnea Index (AHI) >15 at baseline
* Body mass index (BMI) > 35 at baseline
* Severe respiratory disorders (asthma, Chronic obstructive pulmonary disease) at baseline
* Severe cardiovascular disease or severe cardiovascular event < 6 months
* History of stroke or other neurologic chronic illnesses < 6 months
* Have demonstrated impaired mental status
* History of brain tumours, presence of brain metastases or previous cranial irradiation
* Night shift workers
* Excessive lifestyle: massive coffee intake at night, regular excessive cigarette and alcohol consumption in the evening
* Unhealthy sleep hygiene
* Nocturia (the urgent need to urinate more than 2 times during the main sleep period at night) at baseline
* Present diagnosis of depression or psychiatric illness pharmacologically treated
* Diagnosis of insomnia and chronic intake of hypnotic medication at baseline
* Chronic intake of medications that are known to induce sleep disturbance (antihistamines of first generation, cortisone intake > 25 mg/day) or any diagnosed condition that causes known sleep disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: i) Patients with localized, locally advanced or metastatic hormone-sensitive prostate cancer receiving standard of care treatment (including radiotherapy with or without androgen-deprivation treatment (ADT) or ADT alone +/- androgen receptor targeted agent) dependent on disease stage ii) Patients with full-resected early (stage I-III) epithelial BC, ductal carcinoma in situ or lobular carcinoma in situ, without evidence of residual disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
difference in sleep quality | 1 year
  The two groups considered will be group A1, and group A2. This will demonstrate whether there is a difference in sleep quality between these two groups of patients. The difference between time points will establish correlation between treatment initiation and symptom onset, the between group analysis will test whether the link seems to be radiotherapy alone or whether ADT further decreases sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- IOSI, Bellinzona, Switzerland